CLINICAL TRIAL: NCT05651490
Title: RESONATE: A Randomised Controlled Trial of Problem Solving Treatment for Diabetes in Individuals With Poor Diabetes Control
Brief Title: Problem Solving Treatment for Diabetes in Individuals With Poor Diabetes Control
Acronym: RESONATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore Eye Research Institute (Other)
Responsible Party: Principal Investigator, Ecosse Lamoureux, Director, Singapore Eye Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R1596/95/2018
Record Dates: First submitted 2022-12-01; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; problem solving treatment; HbA1c; sugar control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of the two arms: intervention group (PST-D) and attention control group. The random assignment will be based on a code generated by R statistical software, contained within sequential sealed envelopes. The random number sequence will be password protected and available to a statistician external to the study team who will conduct the randomisation process. The randomisation process is designed to yield an expected assignment ratio of 1:1
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (PST-D) (Experimental): Participants in the intervention group will receive usual care comprising of routine follow-up checks from their hospitals on top of the intervention (PST-D). The intervention consists of one introductory session, up to eight weekly treatment sessions, and three monthly maintenance sessions; these are individual sessions of approximately 30 to 45 minutes each and will be conducted over the phone, video call, or face-to-face depending on the participant's preference.
  Interventions: Behavioral: Problem Solving Treatment for Diabetes
- Attention control group (Active Comparator): The participants in the control group will receive usual care comprising of routine follow-up checks from their hospitals. They will also receive one introductory session and up to eight weekly treatment sessions; these are individual sessions of approximately 30 to 45 minutes each and will be conducted over the phone, video call, or face-to-face depending on the participant's preference.
  Interventions: Behavioral: Attention Control Group

INTERVENTIONS:
Behavioral: Problem Solving Treatment for Diabetes — In the introductory session, the structure of and rationale behind PST-D will be explained. The specialist will work with the participant to develop a problem list related to diabetes self-management and smoking cessation, if applicable.
  During the weekly sessions, the participant will be taught and guided through the seven steps of problem solving:
  1. Clarifying and defining the problem
  2. Setting a realistic goal
  3. Brainstorming multiple solutions
  4. Generating pros and cons for each solution
  5. Evaluating and choosing a preferred solution
  6. Developing a specific action plan to implement the solution
  7. Evaluating outcomes from the previous session.
  Participants will also plan to engage in at least 1 enjoyable activity daily during the week.
  The number of sessions will differ based on the specialist's assessment of the participant's problem-solving skills.
  Maintenance sessions will be delivered monthly across 3 months in order to follow-up with participants.
  Arms: Intervention Group (PST-D)
Behavioral: Attention Control Group — During the sessions, the healthcare practitioners will provide general information and recommendations on general health topics such as oral health, hearing loss, sleep, dementia, adult vaccination, influenza, and dengue fever. Participants will also be given handouts adapted from government agencies and/or public bodies, such as HealthHub, National Health Service, National Addictions Management Service, and National Environmental Agency, on these topics. The healthcare practitioners will avoid discussing topics related to diabetes, diet, physical activity, and medication.
  Arms: Attention control group

SUMMARY:
The goal of this randomised controlled trial is to test a cognitive-behavioural intervention, Problem Solving Treatment for Diabetes (PST-D) in patients with type 2 diabetes. The main questions it aims to answer are:

* To evaluate the clinical effectiveness of PST-D compared with the attention control group.
* To determine the impact of PST-D on patient-centred, behavioural, and psychosocial outcomes.
* To identify independent factors associated with an improvement in HbA1c and reductions in incidence and progression diabetic retinopathy, diabetic neuropathy, diabetic peripheral neuropathy, and visual impairment at 18-month follow-up in both groups; and determine if these factors mediate the associations between the PST-D intervention with the above outcomes.
* To quantify the incremental cost-effectiveness of PST-D compared with the attention control group at 18-month follow-up.
* To understand participants' views, experiences, and opinions about PST-D; and the barriers and facilitators to program completion.

Participants will complete blood tests, ocular examinations, and a series of questionnaires at baseline, 6-month, 12-month, and 18-month follow-up. Participants will also complete the intervention/ control group sessions conducted over the phone, video call, or face-to-face depending on the participant's preference.

Researchers will compare the intervention group against the attention control group to determine the effectiveness of PST-D on improving clinical, patient-centred, behavioural, and psychosocial outcomes.

DETAILED DESCRIPTION:
Assuming the recent rise in obesity prevalence persists, the lifetime risk of diabetes in Singapore will almost double by 2050. Poorly controlled diabetes leads to various diabetes-related complications which may consequently require costly lifelong treatment and have a profound impact on patients' quality of life.

Based on a previous trial on problem solving therapy in people with diabetic retinopathy and significant levels of distress, the investigators have designed a cognitive-behavioural intervention which aims to teach individuals skills to cope with and solve problems related to diabetes self-management. This novel intervention will be carried out at one tertiary hospital in Singapore, with the option for interested community-dwelling individuals with diabetes to participate, to facilitate its implementation and transition to the real world setting to assist patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes and at least 1 recent reading of suboptimal glycaemic control (HbA1c ≥7.0%)
* Able to speak English and/or Mandarin
* Singapore citizens or those with Singapore permanent residency status
* Aged 21 years and above
* No cognitive impairment, as assessed using the 6-item Cognitive Impairment Test (6CIT)
* Adequate hearing with/without hearing aids to respond to normal conversation
* Consent to participate in the sessions if randomised to the PST-D treatment arm

Exclusion Criteria:

* Have hearing or cognitive impairment compromising consent or study procedures
* All recent HbA1c readings are <7.0%
* Uncontactable or unwilling/unable to participate in all the PST-D sessions if randomised to the PST-D group

Ages: 21 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c over 18 months | Baseline, 6-month, 12-month, 18-month
  Blood test

SECONDARY OUTCOMES:
Change in total cholesterol, high-density lipoprotein, low-density lipoprotein, triglycerides over 18 months | Baseline, 6-month, 12-month, 18-month
  Blood tests
Incidence and progression of diabetic retinopathy | Baseline, 6-month, 12-month, 18-month
  Grading of digital retinal photographs and spectral-domain optical coherence tomography scans
Incidence and progression of diabetic nephropathy | Baseline, 6-month, 12-month, 18-month
  Blood tests results of epidermal growth factor receptor from serum creatinine and estimated using the CKD-EPI equation
Incidence and progression of diabetic peripheral neuropathy | Baseline, 6-month, 12-month, 18-month
  Semmes-Weinstein monofilament examination (SWME) results
Incidence and progression of distance visual impairment | Baseline, 6-month, 12-month, 18-month
  Pinhole visual acuity values
Change in diabetes self-efficacy over 18 months | Baseline, 6-month, 12-month, 18-month
  Perceived Diabetes Self-management scale.
  Minimum value: 8 Maximum value: 40
  Higher scores indicate more confidence in self-managing one's diabetes.
Change in problem-focused coping self-efficacy over 18 months | Baseline, 6-month, 12-month, 18-month
  Problem-Focusing subscale from Coping Self-Efficacy Scale
  Minimum value: 0 Maximum value: 120
  Higher scores indicate higher level of problem-focused coping self-efficacy.
Change in diabetes self-care activities over 18 months | Baseline, 6-month, 12-month, 18-month
  Diabetes Self-management Questionnaire
  Minimum value: 0 Maximum value: 12
  Higher values indicate more effective self-care.
Change in medication taking behaviour over 18 months | Baseline, 6-month, 12-month, 18-month
  Domains of Subjective Extent of Nonadherence
  It comprises two domains - the extent of and reasons for medication non-adherence over the past 7 days.
  For the Extent of Non-Adherence domain, the overall score is calculated by the average score of the three items, with higher scores indicating greater levels of non-adherence (Minimum value: 0; Maximum value: 4).
  There are 18 items in the Reasons for Non-Adherence domain which stand on their own as descriptors. The reasons scale is a causal indicator model and higher scores indicate greater endorsement of each reason for non-adherence (Minimum value: 0; Maximum value: 4).
Change in diabetes-related quality of life over 18 months | Baseline, 6-month, 12-month, 18-month
  Asian Diabetes Quality of Life
  Minimum value: 18 (English version); 15 (Chinese version) Maximum value: 105 (English version); 90 (Chinese version)
  Higher scores indicate better quality of life.
Cost-effectiveness of PST-D | Baseline, 6-month, 12-month, 18-month
  EQ-5D-5L
  There are five dimensions in the EQ-5D-5L descriptive system - mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Responses to the five dimensions are used to calculate an index score ranging from -0.59 for the worst health state to 1.00 for perfect health. A score of 0 represents death and a negative score indicates a state worse than death.

CONTACTS AND LOCATIONS:
Overall Officials: Ecosse Lamoureux, PhD, Principal Investigator — Singapore Eye Research Institute
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided